CLINICAL TRIAL: NCT03006614
Title: Using PERS(PErsonalized Regimen Selection) Genetic Model Assistant Decision-making System of Neoadjuvant Chemotherapy for Breast Cancer Multicentric, Prospective, Randomized Controlled Phase III Clinical Study
Brief Title: PERS Genetic Model Assistant Decision-making System of Neoadjuvant Chemotherapy for Breast Cancer
Acronym: PERS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Yanxia (Other)
Responsible Party: Sponsor-Investigator, Shi Yanxia, Principal Investigator, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-FXY-077-内科
Record Dates: First submitted 2016-04-28; First posted 2016-12-30 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer Model; Effects of Chemotherapy; Breast Cancer
Keywords: Breast Cancer Model; Effects of Chemotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Epirubicin; Cisplatin; Capecitabine; Gemcitabine; Protons; Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PERS:NVB,DDP,GEM,CAP,H etc. (Experimental): vinorelbine 25mg/m2 d1,d8 iv,q3w cisplatin 70mg/m2 d1，q3w gemcitabine 1000mg/m2 d1,d8,q3w capecitabine 1000mg/m2,bid,d1-14,q3w Trastuzumab
  Interventions: Drug: NVB; Drug: DDP; Drug: CAP; Drug: GEM; Drug: H
- EPI+CTX-T+/-H (Active Comparator): Epirubicin 90mg/m2 d1+ CTX 600mg/m2 d1 q2w, Docetaxel 75mg/m2 +/-herceptin d1,q3w
  Interventions: Drug: EPI; Drug: H; Drug: CTX; Drug: T

INTERVENTIONS:
Drug: NVB
  Other Names: vinorelbine
  Arms: PERS:NVB,DDP,GEM,CAP,H etc.
Drug: EPI
  Other Names: epirubicin
  Arms: EPI+CTX-T+/-H
Drug: DDP
  Other Names: cisplatin
  Arms: PERS:NVB,DDP,GEM,CAP,H etc.
Drug: CAP
  Other Names: capecitabine
  Arms: PERS:NVB,DDP,GEM,CAP,H etc.
Drug: GEM
  Other Names: gemcitabine
  Arms: PERS:NVB,DDP,GEM,CAP,H etc.
Drug: H
  Other Names: Trastuzumab
Drug: CTX
  Other Names: cyclophosphamidem
  Arms: EPI+CTX-T+/-H
Drug: T
  Other Names: docetaxel
  Arms: EPI+CTX-T+/-H

SUMMARY:
This study aims to explore new PERS prediction model can improve the pathological complete response rate of neoadjuvant chemotherapy of breast cancer and disease-free survival.

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized phase III clinical trial. Planning 320 cases.

This study will be divided into two stages. Phase one, 120 cases of local advanced breast cancer (LABC)who need neoadjuvant chemotherapy. Gene prediction model test(PERS) is performed before treatment(ddEC-T+/-H), verify the prediction efficacy of PERS.

Phase two, 200 cases of LABC primary resistant of antharcycline and taxans. Patients were randomized to Arm ddEC-T+/-H and Arm PERS (regimens according to PERS,eg NVB+DDP,capacitabine,gemcitabine and so on) pCR rate and DFS is observed.

ELIGIBILITY:
Inclusion criteria: all of the patients in the trial need to meet

* age: at least 18 years old;
* ECOG(Eastern Cooperative Oncology Group) scoring ≤1;
* confirmed by histology or cytology breast infiltrating ductal carcinoma
* agreed to breast cancer tissue biopsy
* here is a new adjuvant chemotherapy against patients with stage II/III
* According to RECIST criteria, target lesion in patients with at least one, at least one single diameter measurable lesions .Is defined as a measurable lesions with the following method can accurately measure at least one of the diameter of the lesion: lesions or greater diameter 20 mm or measured in conventional methods spiral CT measurement lesions 10 mm diameter or greater. Positron emission tomography (CT) and ultrasound can not be used as measurement method lesions.
* The normal numerical laboratory： The patient's level of organ function must meet the following requirements: enough reserves: bone marrow neutrophils (cent leaves and ribbon neutrophils) absolute count (ANC) ≥1.5*109 / L, or platelets≥ 100*109 / L, or acuity ≥ 9 g/dL and hemoglobin.Liver: bilirubin < 1.5 times the upper limit of normal, alkaline phosphatase (AP), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3.0 times the upper limit of normal (If allowed to AP with liver metastasis, AST, ALT < 5 times the upper limit of normal).Kidney： creatinine clearance or 45 mL/min.
* Signed informed consent;
* is expected to survival in patients with 3 or more months.
* patient adherence and geographic location of residence meet the needs of the follow-up.
* in the research into the group of 7 days before the serum or urine pregnancy test must be negative, and must be for the nursing of patients.Or sterilization surgery, patients after menopause, or agreed to in the research during the treatment and research within 6 months after the end of the treatment period using an approved by the medical contraception (such as intrauterine device (IUD), pill or condoms)

Exclusion Criteria:

* ECOG(Eastern Cooperative Oncology Group) scoring ≥2 ;
* At the same time to accept any other anti-tumor treatment.
* In the past 12 months have congestive heart failure, drug treatment can't control history of arrhythmia, myocardial infarction, etc;
* The serious, which has not been controlled intercurrent infection, organ dysfunction, or serious metabolic disorder of patients;
* Active infection (decided by the researchers.
* According to the researcher's judgment, there is serious to endanger the safety of patients, or patients completed the research associated with disease.
* Pregnancy or breast-feeding women.
* Always have a clear history of neurological or psychiatric disorders, including epilepsy, or dementia.
* A history of other tumors or combined with other tumor patients.
* Before study enrollment for any reason within 30 days of use had not been approved by the local drug ；
* Unwilling or unable to continue to comply with the experimental program, or can not cope with patients follow-up;
* Researchers think that is unfavorable to the participants.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Surgical specimens of breast primary tumors and axillary lymph nodes as measured by Pathological examination. | up to 96 months
  pCR(pathologic complete response)

SECONDARY OUTCOMES:
Time as a measure from randomization to disease recurrence or patients died due to disease progression. | up to 96 months
  DFS(Disease-free survival)

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI(National Cancer Institude) CTC (Clinical Trials Center)v3.0 | up to 96 months
  Safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: YanXia Shi, doctor, Principal Investigator — Sun Yat-sen university of cancer center Recruiting
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No